CLINICAL TRIAL: NCT03202641
Title: Open Lung Strategy, Gas Distribution and Right Heart Function in ARDS Patients: an Open Lung is a Better Heart
Brief Title: Open Lung Strategy, Gas Distribution and Right Heart Function in ARDS Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLA-HEART
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ARDS, Human; Lung Injury, Acute; Respiratory Distress Syndrome; Mechanical Ventilation Complication; Alveolar Edema; Right Heart Failure; Right Ventricular Dysfunction
Keywords: ARDS; PEEP titration; Open Lung Strategy; Right heart function; Lung recruitment maneuver; Esophageal Pressure; Respiratory system compliance
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Heart Failure; Ventricular Dysfunction, Right

STUDY DESIGN:
Intervention Model Description: Physiologic crossover study. There is no randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP_titration (Experimental): There is no randomization in this interventional, crossover, physiological study. All participants will receive the same procedures in the same order. The investigators will compare two PEEPs ("PEEPARDSnet" vs. "PEEPLRM").
  Interventions:
  1. PEEP ARDSnet: we will select the PEEP based on low PEEP/high FiO2 table (ARDSnet).
  2. PEEP LRM: we will perform a lung recruitment maneuver (LRM) and select PEEP based on transpulmonary pressure.
  Interventions: Procedure: PEEP ARDSnet; Procedure: PEEP LRM

INTERVENTIONS:
Procedure: PEEP ARDSnet — PEEP settings based on the low PEEP/high FiO2 table
Procedure: PEEP LRM — A lung recruitment maneuver (LRM) followed by PEEP guided by transpulmonary pressure.

SUMMARY:
The goal of this interventional crossover study, in intubated and mechanically ventilated Acute Respiratory Distress Syndrome (ARDS) patients, is to compare two positive end-expiratory pressure (PEEP) titration techniques regarding: respiratory mechanics, gas exchange, changes in aeration, ventilation/perfusion matching its impact on cardiac function, especially the right heart (RH). The PEEP titration techniques are: PEEP selection based on low PEEP/high FiO2 table ("PEEPARDSnet") and lung recruitment maneuver (LRM) plus PEEPdec titration based on the best compliance of the respiratory system("PEEPLRM").

DETAILED DESCRIPTION:
A recent large observational study published on JAMA showed that Acute Respiratory Distress Syndrome (ARDS) is associated with high mortality and developed in 10.4% of 29,144 patients admitted to the intensive care unit from 50 countries across 5 continents. Mechanical ventilation is the cornerstone for lung treatment during ARDS. Lung protective ventilation improved ARDS outcome significantly. However, it is still unclear what method should be used to select levels of positive end-expiratory pressure (PEEP).

In the current study proposal, the investigators hypothesized that, when ARDS lungs are recruitable, a lung recruitment maneuver (LRM) and PEEP titration ("PEEPLRM") improve ventilation/perfusion matching and decreased right heart workload when compared to the actual standard of care PEEP selection based on low PEEP/high FiO2 table ("PEEPARDSnet").

The investigators will test this hypothesis in an interventional crossover study.

50 patients with ARDS will be enrolled in a physiological and lung and heart imaging study.

The protocol is divided in the following phases:

A) "PEEPARDSnet": setting PEEP according to the ARDSnet table (low PEEP/ high FiO2)

B) Recruitability assessment sequence:

P-V curve tool (Hamilton ventilator): evaluate patient recruitability, among three criteria, two must be positive to consider a subject recruitable: (1) Presence of a lower inflection point (2) Linear compliance measured more than 2 times higher than the dynamic compliance (3) Increase in volume of more than 300mL during the descendant limb of the PV curve at a same given pressure (20 cmH2O)(Hysteresis property).

C)"PEEPLRM": LRM plus PEEP decremental trial guided by best compliance. Lung and heart response to "PEEPLRM": we will compare the driving pressure (DP) value (DP = Plateau pressure - PEEP) and transthoracic echocardiography (TTE) with the values at PEEPARDSnet. In the advent of an increased DP and/or new onset of abnormal values at the TTE, we will resume the PEEPARDSnet settings during the 48h follow-up phase.

Before and after the lung recruitment maneuver and decremental PEEP trial, we will collect:

1. Respiratory system mechanics
2. Lung volumes
3. Gas exchange
4. Hemodynamic parameters
5. Electrical Impedance Tomography (EIT) ventilation and perfusion data
6. Transthoracic echocardiographic indices of RH function

Follow-up phase:

In 24 and 48 hours, if the subject did not present a negative response to "PEEPLRM" as described above , we will repeat the recruitment maneuver and the decremental PEEP trial and and we will collect:

1. Respiratory system mechanics (i.e. driving pressure)
2. Lung volumes
3. Gas exchange
4. Hemodynamic parameters
5. EIT ventilation and perfusion data
6. Transthoracic echocardiographic indices of RH function

before and after the aforementioned intervention.

ELIGIBILITY:
Inclusion Criteria:

* ARDS diagnosis within 72h after intubation
* Severe to moderate ARDS (PaO2 / FiO2 < 200 mmHg) with PEEP>5 cmH2O
* Presence of an arterial line
* Between 18 and 85 years old

Exclusion Criteria:

* Persistent systolic blood pressure < 90 mmHg and/or >180 mmHg despite the use of vasopressor or vasodilators
* Increment in vasopressors over the past two hour just before enrollment of: more than 15 mcg/min for norepinephrine and dopamine, more than 10 mcg/min in epinephrine; and more than 50 mcg/ min for phenylephrine.
* Advanced lung disease confirmed by computed tomography findings
* Presence or history of pneumothorax
* Severe coagulopathy (INR ≥ 4)
* Severe thrombocytopenia (Platelets count ≤ 5,000/mm3)
* Usage of any devices with electric current generation such as pacemaker or internal cardiac defibrillator
* Recent esophageal trauma or surgery
* Known presence of esophageal varices
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Driving Pressure (cmH2O) | 1h (Phase A: "PEEP ARDSnet") and 2h (Phase C: "PEEP LRM") after the beginning of the study procedures
  The primary endpoint of this study is to describe the airways driving pressures (defined as Plateau Pressure minus PEEP) during "PEEP ARDSnet" and "PEEP LRM".

OTHER OUTCOMES:
Chest wall and lung elastances (cmH2O/L) | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  This exploratory outcome represents the respiratory system elastance. The respiratory system elastance (ERS = EL + ECW) is the sum of lung elastance (EL) and chest wall (ECW) elastance. In order to measure ERS, we will need airway pressure (measured by connecting the endotracheal tube with a pressure transducer) and pleural pressure (measured by placing an esophageal balloon connected to a pressure transducer, the esophageal pressure is a surrogate of the pleural pressure).
Dead space (%) | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  This exploratory outcome is the volume (as a percent) of a breath that does not participate in gas exchange.The measure will be made using infrared absorption technology by a mainstream analyzer positioned distally to the Y piece and connected to a capnogram.
Right heart function (Transthoracic Echocardiography) | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  Exploratory outcome
Gas distribution, gas content, end-expiratory lung volume (using Electrical Impedance Tomography) | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  Exploratory outcome
Ventilation/perfusion matching (using Electrical Impedance Tomography) | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  Exploratory outcome
Blood arterial and central venous pressures | 1h (Phase A: "PEEP ARDSnet"), 2h (Phase C: "PEEP LRM"), 24h and 48h after the beginning of the study procedures
  Exploratory outcome
Days free of mechanical ventilation | 28 days
  Exploratory outcome
ICU length of stay | 28 days
  Exploratory outcome
Hospital length of stay | 28 days
  Exploratory outcome
Mortality | 28 days
  Exploratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, RRT, PhD, Principal Investigator — Massachusetts General Hospital; Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital; Roberta De Santis Santiago, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachussets General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashbaugh DG, Bigelow DB, Petty TL, Levine BE. Acute respiratory distress in adults. Lancet. 1967 Aug 12;2(7511):319-23. doi: 10.1016/s0140-6736(67)90168-7. No abstract available. PMID 4143721
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Lachmann B. Open Lung in ARDS. Minerva Anestesiol. 2002 Sep;68(9):637-42; discussion 640, 643. No abstract available. PMID 12370679
- [Background] Kacmarek RM, Villar J, Sulemanji D, Montiel R, Ferrando C, Blanco J, Koh Y, Soler JA, Martinez D, Hernandez M, Tucci M, Borges JB, Lubillo S, Santos A, Araujo JB, Amato MB, Suarez-Sipmann F; Open Lung Approach Network. Open Lung Approach for the Acute Respiratory Distress Syndrome: A Pilot, Randomized Controlled Trial. Crit Care Med. 2016 Jan;44(1):32-42. doi: 10.1097/CCM.0000000000001383. PMID 26672923
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2014 Mar 6;370(10):980. doi: 10.1056/NEJMc1400293. No abstract available. PMID 24597883
- [Background] Borges JB, Okamoto VN, Matos GF, Caramez MP, Arantes PR, Barros F, Souza CE, Victorino JA, Kacmarek RM, Barbas CS, Carvalho CR, Amato MB. Reversibility of lung collapse and hypoxemia in early acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Aug 1;174(3):268-78. doi: 10.1164/rccm.200506-976OC. Epub 2006 May 11. PMID 16690982
- [Background] de Matos GF, Stanzani F, Passos RH, Fontana MF, Albaladejo R, Caserta RE, Santos DC, Borges JB, Amato MB, Barbas CS. How large is the lung recruitability in early acute respiratory distress syndrome: a prospective case series of patients monitored by computed tomography. Crit Care. 2012 Jan 8;16(1):R4. doi: 10.1186/cc10602. PMID 22226331
- [Background] Pirrone M, Fisher D, Chipman D, Imber DA, Corona J, Mietto C, Kacmarek RM, Berra L. Recruitment Maneuvers and Positive End-Expiratory Pressure Titration in Morbidly Obese ICU Patients. Crit Care Med. 2016 Feb;44(2):300-7. doi: 10.1097/CCM.0000000000001387. PMID 26584196
- [Background] Fumagalli J, Berra L, Zhang C, Pirrone M, Santiago RRS, Gomes S, Magni F, Dos Santos GAB, Bennett D, Torsani V, Fisher D, Morais C, Amato MBP, Kacmarek RM. Transpulmonary Pressure Describes Lung Morphology During Decremental Positive End-Expiratory Pressure Trials in Obesity. Crit Care Med. 2017 Aug;45(8):1374-1381. doi: 10.1097/CCM.0000000000002460. PMID 28708679
- [Background] Pinsky MR. My paper 20 years later: Effect of positive end-expiratory pressure on right ventricular function in humans. Intensive Care Med. 2014 Jul;40(7):935-41. doi: 10.1007/s00134-014-3294-8. Epub 2014 Apr 24. PMID 24760121
- [Background] Lansdorp B, Hofhuizen C, van Lavieren M, van Swieten H, Lemson J, van Putten MJ, van der Hoeven JG, Pickkers P. Mechanical ventilation-induced intrathoracic pressure distribution and heart-lung interactions*. Crit Care Med. 2014 Sep;42(9):1983-90. doi: 10.1097/CCM.0000000000000345. PMID 24743042
- [Background] Matamis D, Lemaire F, Harf A, Brun-Buisson C, Ansquer JC, Atlan G. Total respiratory pressure-volume curves in the adult respiratory distress syndrome. Chest. 1984 Jul;86(1):58-66. doi: 10.1378/chest.86.1.58. PMID 6734293
- [Background] Demory D, Arnal JM, Wysocki M, Donati S, Granier I, Corno G, Durand-Gasselin J. Recruitability of the lung estimated by the pressure volume curve hysteresis in ARDS patients. Intensive Care Med. 2008 Nov;34(11):2019-25. doi: 10.1007/s00134-008-1167-8. Epub 2008 Jun 25. PMID 18575846
- [Background] Maggiore SM, Jonson B, Richard JC, Jaber S, Lemaire F, Brochard L. Alveolar derecruitment at decremental positive end-expiratory pressure levels in acute lung injury: comparison with the lower inflection point, oxygenation, and compliance. Am J Respir Crit Care Med. 2001 Sep 1;164(5):795-801. doi: 10.1164/ajrccm.164.5.2006071. PMID 11549535
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507